CLINICAL TRIAL: NCT02781077
Title: Intensity of a Task-Oriented Exercise Program for Optimizing Walking Competency in Stroke Survivors
Brief Title: Intensity of Task-Oriented Exercises
Acronym: TOE
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Thin Thin Moe, Ph D candidate, Mahidol University
Other Study IDs: 2-2016
Record Dates: First submitted 2016-05-16; First posted 2016-05-24 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Stroke
Keywords: Stroke; walking competency; Task-oriented exercise program; Exercise intensity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Structured, Progressive, Task-oriented exercise program — The intervention is walking related task-oriented exercise program with three progressive steps at moderate to high intensity. Each step consists of 60 minutes last ten tasks to optimize walking function of stroke individuals.

SUMMARY:
In an observational study, the energy consumption of stroke individuals during performing the structured, progressive task-oriented exercise program for walking rehabilitation will be measured in order to confirm the intensity demand in the range of moderate to vigorous.

DETAILED DESCRIPTION:
Community reintegration is often significantly affected in the majority of stroke individuals. To fulfill the requirements of a proper home exercise program in walking rehabilitation for stroke victims, investigators structured the task-oriented exercise program with minimal supervision. This exercise program is structured with challenging walking-related activities based on motor learning principle and Gentile's progression of the motor task. The strengthening and balance components, aerobic conditioning and walking adaptability are composed of an exercise program to optimize walking ability. There are sixty minutes last ten exercises in each three progression steps of this exercise program. For the training effect to occur, each step of exercise program is designed by increasing demand of intensity in the range from moderate to vigorous. To confirming progressive energy demand, the purpose of this study is to investigate the intensity demand of three steps task- oriented home exercise program on walking competency in individual post stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Either side of both type first stroke with confirmatory diagnosis by CT Scan and MRI.
2. Age above 20 years old.
3. Moderate severity of stroke measured by the modified Rankin Scale (mRS- 3)
4. Able to comprehend the instructions with good cognition measured by Mini-Mental State Examination (MMSE > 23).

Exclusion Criteria:

1. Diagnosed with other neurological disorder such as Parkinson's disease, peripheral nerve injury.
2. Serious cardiac conditions (angina and myocardial infarction during the previous month, resting heart rate of more than 120, a systolic blood pressure of more than 180 mm Hg, and a diastolic blood pressure of more than 100 mm Hg)
3. Fugl Meyer Assessment score (lower extremity) less than ≤ 21
4. Significant hip, knee and ankle contracture that would limit ambulation (Fugl Meyer (ROM) ≤1 in each joint).
5. Orthopedic and rheumatological disorder with weight bearing pain (Fugl Meyer (pain) ≤ 1 in hip, knee and ankle joint movement).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke individuals who able to walk without physical assistance.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of Oxygen Consumption (VO2rate) (ml/kg/min) | 1 week
  The amount of oxygen consumption of participants will be measured by using Oxycon Mobile spirometer (OM) on 3 occasions: during performing step I,II and III of exercise program with 1-2 days apart between each step.

SECONDARY OUTCOMES:
Heart Rate | 1 week
  Heart rate of participants will be measured on 3 occasions: during performing step I,II and III of exercise program with 1-2 days apart between each step
Metabolic Equivalents (METs) [VO2max (ml.kg-1.m-1)/VO2rest(ml.kg-1.m-1)] | 1 week
  METs is a way to express the energy cost of activity, calculated by using the formula of VO2/VO2rest on 3 occasions:during performing step I,II and III of exercise program with 1-2 days apart between each step.
Borg Rating of Perceived Exertion scale (RPE) | 1 week
  The feeling of how strenuous a given exercise to a patient related to the amount of effort exerted is rated by the categorical-ratio scale of 0 to 10 RPE on 3 occasions: during performing step I,II and III of exercise program with 1-2 days apart between each step.

CONTACTS AND LOCATIONS:
Overall Officials: Thin Thin Moe, M.Med.Tech, Principal Investigator — Mahidol University; Chutima Jalayondeja, Dr.P.H. MSc, Study Chair — Mahidol University; Sopa Pichaiyongwongdee, M.Sc. B.Sc, Study Director — Mahidol University; Vimonwan Hiengkaew, PhD. MSc, Study Director — Mahidol University; Jarugool Tretriluxana, PhD. MSc, Study Director — Mahidol University
Locations (1):
- Mahidol University, Bangkok, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided